CLINICAL TRIAL: NCT02846337
Title: Ultrafiltration Versus Medical Therapies in the Management of the Cardio Renal Syndrome
Acronym: UF-CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL15_0077; 2016-A00518-43 (Other: ID-RCB)
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Cardio-renal Syndrome
Keywords: cardio-renal syndrome; hemodialysis; peritoneal dialysis; hemofiltration; composite endpoint
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ULTRAFILTRATION (Experimental): The ultrafiltration sodium-overload extraction will be chosen by the patient nephrologist and the patient himself (according to his comorbidities) among the following one: peritoneal dialysis (at least a daily contact), hemodialysis (>1 session per week) or isolated ultrafiltration (>1 session per week). Ultrafiltration technique could change throughout the care
  Interventions: Procedure: ULTRAFILTRATION
- ENHANCED MEDICAL TREATMENT (Other): The control group called "enhanced medical treatment" will not benefit of ultrafiltration (except refractory pulmonary edema, or terminal kidney failure requiring extra renal depuration). These situations will not be considered as protocol violation, because they are scientifically indicated for extra renal depuration.
  Interventions: Procedure: ENHANCED MEDICAL TREATMENT

INTERVENTIONS:
Procedure: ULTRAFILTRATION — Peritoneal dialysis: at least one daily contact, 5 days a week minimum, with a hypertonic solution. Le number of contact et the stasis duration will be decided by the practitioner.
  Hemodialysis: at least one hemodialysis per week, one hemofiltration and/or hemodiafiltration per week, and at least 2 liter of ultrafiltrate extraction per week. In case of serious interdialytic weight gain, and/or hemodynamic unsteadiness, sessions can be up to 6 per weeks. Sessions duration will be adjusted to the needful ultrafiltrate and hemodynamic tolerance.
  Isolated ultrafiltration: at least once a week, and includes an extraction of minimum 2 liter ultrafiltrate in less than 4 hours. It could be done, according to routines and department capacity, on a hemodialysis generator, plasmatic exchange generator, or mobile ultrafiltration device.
  Arms: ULTRAFILTRATION
Procedure: ENHANCED MEDICAL TREATMENT — * Close cardiologic and nephrologic follow-up, minimum 4 times a year, This incidence matches the heart failure, and chronic kidney failure care guidance for our sample
  * Medical care adjustment in order to apply European and American guidance for chronic heart failure care
  * Hydric, caloric, peptic and sodium input evaluation by a dietician, and adjustment if needed
  * Physical rehabilitation suggestions by a physiologist
  * Evaluation of an interventional approach requirement, and implementation if needed (pacemaker, defibrillator, cardiac resynchronization, diagnosis and therapeutic coronary angiography, ventricular stimulator) according to European and American guidance.
  Arms: ENHANCED MEDICAL TREATMENT

SUMMARY:
Type 2 cardio renal syndrome is defined by the occurrence or the exacerbation of a kidney failure induced by a chronic heart failure. Sodium overload is one of the main causes leading to the occurrence or the exacerbation of this syndrome. Some patients have a massive sodium retention on which medications are not effective enough. These patients have no further therapeutic options because of the refractory congestion and a 3-months mortality rate around 15%, frequent rehospitalization (3-months rehospitalization rate at 71%) and an excessively impaired quality of life.

For those refractory heart failure with cardio renal syndrome, nephrology departments resort to non-medication sodium extraction (hemodialysis, peritoneal dialysis, isolated ultrafiltration). Between 2002 and 2008, 927 French patients would have start dialysis in this situation. In 2013, 174 patients start dialysis in 97 dialysis centers. French National Authority of Health recently published new Good Practice Guidance thereupon, strengthened by the increasing number of publications and the widespread use of this technique. There is therefore a consensus among professionals about the benefits of such a technique in those indications. However, bibliographical data are not strong enough to support a strong level of evidence. None of foresight strategies have been compared to others in a proper randomized controlled trial, and there is no clue about any suspected superiority from one strategy to another.

So far, the investigators propound invasive, expensive and not validated techniques to patients with functional and vital prognosis altered. The investigators think it's essential to prove the efficacy of such an approach. They wish to quantify those techniques impact on rehospitalization, with a consideration for the potential survival impact.

It seems unethical to evaluate separated techniques, taking in account that patients with severe heart failure will switch from one technique to another among their care. It is therefore crucial to validate benefits from an invasive procedure (hemodialysis, peritoneal dialysis, isolated ultrafiltration) compared to a medication-restricted care.

ELIGIBILITY:
Inclusion Criteria:

* Severe heart failure with recurring congestive symptoms and at least one the following criteria :

  * At least 2 hospitalization > 24 hours for congestive symptoms among the 12 months before the inclusion, whose latest one was in the 6 months before the inclusion
  * Persistent congestive symptoms throughout 30 days (case history) before the randomization: dyspnea NYHA III or IV, lower limbs edema and/or ascites.
* Diuretic treatment with at least 250mg furosemide per day (or 6mg bumetanide)during at least 1 month
* Cardiac medical treatment enhanced by the European cardiology society guidance (except intolerance, and/or contraindication) and according to patient cardiologist.
* Non terminal kidney disease or failure : estimated glomerular filtration rate (GFR) (CKD-Epi formula) between 20 and 90 mL/min/1.73m² (or GFR estimated between 60 and 90 mL/min/1.73m² with proteinuria and/or hematuria) and urea rate under 50mmol/L

Exclusion Criteria:

* Cardiogenic shock or situations that contraindicate the ultrafiltration technique elsewhere than shock room
* Patient who already had long course ultrafiltration for more than 3 months, or not available because of end-stage renal failure
* Biventricular pacemaker implementation, single or dual chamber pacemaker implementation, or defibrillator implementation up to 15 days before the inclusion
* Vasoactive drugs ambulatory treatment (dobutamine, dopamine, adrenalin, noradrenalin)
* General condition incompatible with any ultrafiltration techniques
* Age under 18
* Pregnant or lactating women
* Law-protected patients
* Patients that can't submit to the follow-up for geographical, social or mental reasons
* Unwillingness to be treated by ultrafiltration techniques
* Patients who don't belong to the national social security system, or similar system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
death and/or unscheduled hospitalization | up to 12 months post-randomization
  The primary outcome measure is a combined measure including death whatever the cause, and/or unscheduled hospitalization for acute decompensated heart failure. For each groups, deaths, cause and time of deaths will be recorded. Hospitalization date, duration, location, and reason will be recorded. The "hospitalization" setting and the "acute decompensated heart failure" setting will be endorsed by an event validation committee.

SECONDARY OUTCOMES:
Survival | 12 months
  number of days spent alive and not hospitalized
Survival | 12 months
  Intervention effect on one-year overall survival
Hospitalization for acute decompensated heart failure | up to 12 months post- randomization
  Intervention effect on :
  * Period before first unscheduled hospitalization for acute decompensated heart failure
  * Number and duration of hospitalizations for acute heart failure (scheduled or not) throughout the year
  * Number and duration of unscheduled hospitalization for acute heart failure throughout the year.
Change in NYHA classification | randomization day and 12 months post randomization.
  New York Health Association - Measurement scale to classify heart failure in 4 stages (stage 1 ; no symptoms)
Change in 6MWT - Six-Minute Walk Test | randomization day and 12 months post randomization.
  Six-minute walk test with an experimented physiologist. The distance in meters is retained.
Change in MLwHF form | randomization day and 12 months post randomization.
  Minnesota Living with Heart Failure - Quality of life self-administered survey focusing on heart failure symptoms (21 items with 1 : slightly to 5 : al lot) Safety issue? 0 Yes 1 No
Change in SF36 form | randomization day and 12 months post randomization.
  Short Form 36 : Quality of life self-administered survey with 36 items about 8 dimensions including a physical and mental score.
Death occurrence attributable to ultrafiltration technique | up to 12 months post- randomization
  Safety: Death occurrence attributable to ultrafiltration technique, validated by an independent supervisory board, and any adverse event.
Change in Brain Natriuretic Peptide and/or NT-Probating Natriuretic Peptide rate | randomization day and 12 months post randomization
  Following biological features variation : Brain Natriuretic Peptide (BNP) and/or NT-ProBNP
Change in total bilirubin rate | randomization day, then 3, 6 and 12 months post randomization
  Following biological features variation : total bilirubin
Change high-sensitivity T troponin rate | randomization day and 12 months post randomization
  Following biological features variation : high-sensitivity T troponin
Change in hemoglobin rate | randomization day and 12 months post randomization
  Following biological features variation : hemoglobin
Change in Left ventricular ejection fraction (LVEF) | randomization day and 12 months post randomization
  Following echocardiographic parameters features : left systolic function (LVEF)
Change in Tricuspid annular plane systolic excursion (TAPSE) | randomization day and 12 months post randomization
  Following echocardiographic parameters features :right systolic function (TAPSE)
Change in tricuspid annular velocity | randomization day and 12 months post randomization
  Following echocardiographic parameters features : right systolic function assessed by tricuspid annular velocity measured with Pulsed Doppler tissue imaging
Change in transmitral patterns classification | randomization day and 12 months post randomization
  Following echocardiographic parameters features : left diastolic function assessed by transmitral patterns classification
Change in E/E' ratio | randomization day and 12 months post randomization
  Following echocardiographic parameters features : E/E'
Change in pulmonary artery systolic pressure (PASP) | randomization day and 12 months post randomization
  Following echocardiographic parameters features : pulmonary artery systolic pressure (PASP)
Change in Surface of the Left Atrium | randomization day and 12 months post randomization
  Following echocardiographic parameters features : Surface of the Left Atrium
Change in right atrial pressure | randomization day and 12 months post randomization
  Following echocardiographic parameters features : Impact on right ventricular function assessed by right atrial pressure
Change in cardiac index | randomization day and 12 months post randomization
  Following echocardiographic parameters features : cardiac index
Change in cardiac flow | randomization day and 12 months post randomization
  Following echocardiographic parameters features : cardiac flow

CONTACTS AND LOCATIONS:
Overall Officials: Laurent JUILLARD, Principal Investigator — Hospices Civils de Lyon, 69002 LYON France
Locations (1):
- Hospices Civils de Lyon, Hôpital E Herriot, Service de néphrologie, 5 place d'Arsonval, Lyon, Rhones Alpes, France